CLINICAL TRIAL: NCT01312272
Title: Does Acute Oxytocin Administration Enhance Social Cognition in Individuals With Schizophrenia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael C. Davis, M.D., Ph.D., Fellow / Physician, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCC 2011-020223
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Social Intelligence; Perception, Social; Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inactive nasal spray (Placebo Comparator): A placebo nasal spray will be prepared to be otherwise identical to the active treatment nasal spray except lacking oxytocin. The ingredients in the inactive nasal spray are mannitol, glycerin, and preserved water.
  Interventions: Drug: Inactive placebo nasal spray
- Intranasal Oxytocin (Experimental): Oxytocin nasal spray (40 units/ml) will be administered in a single intranasal dose of 40 IU. Its formula is: oxytocin 1 unit/mg mannitol trituration 0.2Gm + glycerin USP 0.1ml + preserved water 5ml.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 40 units/ml nasal spray: use 5 sprays per nostril (40 IU total) one time
  Arms: Intranasal Oxytocin
Drug: Inactive placebo nasal spray — A placebo nasal spray will be prepared identically to the oxytocin nasal spray except lacking oxytocin. Its ingredients are mannitol, glycerin, and preserved water. It will be administered at 5 sprays to each nostril, one time.
  Arms: Inactive nasal spray

SUMMARY:
Individuals with schizophrenia have been found to have deficits in social cognition, which is defined as the functions that are engaged during social interactions. Social cognition has been found to be critical in predicting multiple aspects of community functioning. There are no currently available medications that have been consistently found to improve social cognition in individuals with schizophrenia. Oxytocin functions as a neurotransmitter that is thought to be involved in multiple aspects of social behavior and related emotions. In this study, we test the hypothesis that acute administration of intranasal oxytocin will improve social cognition in individuals with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is characterized by the presence of positive symptoms (delusions, hallucinations, disorganization of thought process and behavior) as well as negative symptoms (blunted affect, alogia, and avolition), neurocognitive deficits, and impaired social cognition. While positive symptoms can often respond well to antipsychotic medications, the latter symptoms are more difficult to treat. In this study, we will focus on social cognition, which is defined as the functions that are engaged during social interactions. Social cognition has been categorized into four main domains: theory of mind, social perception, attributional bias, and emotional processing. Social cognition in patients with schizophrenia has been found to be critical in predicting multiple aspects of community functioning. There are currently two broad approaches to improve social cognition in patients with schizophrenia: pharmacological and psychosocial interventions. While psychosocial interventions (training exercises to target improvement in domains of social cognition) have shown some benefit, their resultant improvements have been limited in their distribution across multiple domains as well as their generalization to improved functioning in the community. Pharmacological trials have yielded mixed results, and there are not any currently available medications that have been consistently found to improve social cognition in patients with schizophrenia2. One potential future therapeutic target for enhancing social cognition is the oxytocin system.

Oxytocin is a nine-amino acid peptide that, in addition to its role in the periphery for regulating lactation and uterine contractions, functions centrally as a neurotransmitter which is involved in multiple aspects of social behavior and related emotions. Specifically, it has been found to modulate emotion recognition, trust, eye contact, empathic accuracy, as well as envy and gloating. Given oxytocin's role in social functioning, in conjunction with the deficits in social functioning found frequently in individuals with schizophrenia, there have been several studies over the past three decades examining the oxytocin system in humans with schizophrenia and in rodent experimental models.

It has been found that individuals with schizophrenia do not show the same level of increase in oxytocin as normal controls in response to trust-related interpersonal interactions, and low plasma oxytocin predicted negative symptoms of schizophrenia. Additionally, it has also been found that plasma oxytocin levels predicted the ability of patients with schizophrenia to identify facial expressions. Finally, it has been found recently that sustained regular administration of intranasal oxytocin significantly reduced both positive and negative symptoms of schizophrenia. Thus, there is significant evidence supporting further research studying the effect of oxytocin on social cognition. It is not yet known if exogenous administration of oxytocin will have acute effects on neuropsychological measures of social cognition in individuals with schizophrenia, and this is the focus of this proposed pilot study.

The overall hypothesis guiding this study is that acute oxytocin administration will improve social cognition (as assessed by a composite score comprising two measures of "low level" social cognitive processes and two measures of "high level" social cognitive processes) in individuals with schizophrenia. Our primary goals are to assess the feasibility of this experimental paradigm and to generate pilot data and obtain estimates of effect sizes which can be used in planning future larger studies.

ELIGIBILITY:
Inclusion Criteria:

* Veteran being treated in the Veterans Administration Healthcare System
* Meet DSM-IV-TR criteria for Schizophrenia
* At least 6 months since any hospitalization or substantial increase in level of care for an acute exacerbation of psychotic symptoms
* At least 1 month since meeting the criteria for having a major depressive episode
* At least 6 months since any behaviors suggesting any potential danger to self or others
* Adherence to the regular administration of an antipsychotic medication (e.g., risperidone, olanzapine, quetiapine, ziprasidone, aripiprazole, paliperidone, iloperidone, asenapine, fluphenazine, haloperidol, loxapine, molindone, perphenazine, thiothixene, chlorpromazine, clozapine)
* Dose of antipsychotic medication not varying by more than 25% over the 3 months prior to study participation
* No acute medical problems
* Chronic medical conditions (e.g., hypertension, diabetes, dyslipidemia) consistently treated and stable for at least 3 months prior to study participation
* Ability to provide signed informed consent and to cooperate with study procedures

Exclusion Criteria:

* Documented history of mental retardation or severe learning disability
* History of treatment with electroconvulsive therapy within 6 months prior to study participation
* History of neurological or neuropsychiatric condition (e.g., stroke, severe traumatic brain injury, epilepsy, etc.)
* Documented history of persistent substance abuse or dependence within 6 months prior to study participation
* History of hyponatremia within the past 6 months
* Allergic rhinitis or other inflammation of the nasal mucosa

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marder, M.D., Principal Investigator — VA Greater Los Angeles
Locations (1):
- West Los Angeles VA Healthcare Center, Los Angeles, California, United States

REFERENCES:
- [Background] Bartz JA, Zaki J, Bolger N, Hollander E, Ludwig NN, Kolevzon A, Ochsner KN. Oxytocin selectively improves empathic accuracy. Psychol Sci. 2010 Oct;21(10):1426-8. doi: 10.1177/0956797610383439. Epub 2010 Sep 20. No abstract available. PMID 20855907
- [Background] Domes G, Heinrichs M, Michel A, Berger C, Herpertz SC. Oxytocin improves "mind-reading" in humans. Biol Psychiatry. 2007 Mar 15;61(6):731-3. doi: 10.1016/j.biopsych.2006.07.015. Epub 2006 Nov 29. PMID 17137561
- [Background] Feifel D, Macdonald K, Nguyen A, Cobb P, Warlan H, Galangue B, Minassian A, Becker O, Cooper J, Perry W, Lefebvre M, Gonzales J, Hadley A. Adjunctive intranasal oxytocin reduces symptoms in schizophrenia patients. Biol Psychiatry. 2010 Oct 1;68(7):678-80. doi: 10.1016/j.biopsych.2010.04.039. Epub 2010 Jul 7. PMID 20615494
- [Background] Goldman M, Marlow-O'Connor M, Torres I, Carter CS. Diminished plasma oxytocin in schizophrenic patients with neuroendocrine dysfunction and emotional deficits. Schizophr Res. 2008 Jan;98(1-3):247-55. doi: 10.1016/j.schres.2007.09.019. Epub 2007 Oct 24. PMID 17961988
- [Background] Guastella AJ, Mitchell PB, Dadds MR. Oxytocin increases gaze to the eye region of human faces. Biol Psychiatry. 2008 Jan 1;63(1):3-5. doi: 10.1016/j.biopsych.2007.06.026. Epub 2007 Sep 21. PMID 17888410
- [Background] Keri S, Kiss I, Kelemen O. Sharing secrets: oxytocin and trust in schizophrenia. Soc Neurosci. 2009;4(4):287-93. doi: 10.1080/17470910802319710. Epub 2008 Aug 1. PMID 18671168
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Shamay-Tsoory SG, Fischer M, Dvash J, Harari H, Perach-Bloom N, Levkovitz Y. Intranasal administration of oxytocin increases envy and schadenfreude (gloating). Biol Psychiatry. 2009 Nov 1;66(9):864-70. doi: 10.1016/j.biopsych.2009.06.009. Epub 2009 Jul 29. PMID 19640508
- [Background] Webber MA, Marder SR. Better pharmacotherapy for schizophrenia: what does the future hold? Curr Psychiatry Rep. 2008 Aug;10(4):352-8. doi: 10.1007/s11920-008-0056-8. PMID 18627675
- [Result] Davis MC, Lee J, Horan WP, Clarke AD, McGee MR, Green MF, Marder SR. Effects of single dose intranasal oxytocin on social cognition in schizophrenia. Schizophr Res. 2013 Jul;147(2-3):393-7. doi: 10.1016/j.schres.2013.04.023. Epub 2013 May 12. PMID 23676253
- See also: Link to PubMed journal article citation for peer-reviewed publication describing study — http://www.ncbi.nlm.nih.gov/pubmed/23676253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.1) | 48.6 (6.6) | 48.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 3 | 1 | 4
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Social Cognition Composite Measure
Description: Our primary outcome measure will be a composite score created by calculating the mean of the four main social cognition measures assessed in this study (two "high-level" measures and two "low-level" measures). Because these measures are not on the same scale, we will first z-score (center and scale) each of the four measures at each time point using the baseline mean and standard deviation of the whole sample and then calculate the mean of the z-scores to create the composite social cognition score.
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: Change in z-score
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
Change in z-score | 0.10 (0.35) | 0.23 (0.36)

2. Secondary Outcome: Theory of Mind Assessment (High Level Social Cognition)
Description: The Awareness of Social Inference Test (TASIT Part III: Social Inference - Enriched) will be administered to assess theory of mind.
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: Change in z-score
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
Change in z-score | -0.01 (0.47) | 0.18 (0.83)

3. Secondary Outcome: Empathy
Description: Empathy was assessed using the Emotional Perspective Taking Task (EPTT) (Derntl et al., 2009). In this task, subjects are presented with 60 digital images depicting two individuals in a social interaction, with one individual's face masked. Subjects are asked to infer the emotional expression of the masked face, selecting between two choices. Scenes portray 5 basic emotions as well as neutrality and each image is displayed for 4 s each.
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: Change in z-score
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
Change in z-score | 0.24 (0.63) | 0.61 (0.76)

4. Secondary Outcome: Social Perception Assessment (Low Level Social Cognition)
Description: We will assess social perception using the Half-Profile of Nonverbal Sensitivity (Half-PONS). Brief scenes are shown that include facial expressions, voice intonations, and/or body gestures. Subjects select a label that best describes the situation. The dependent measure is the total number of correct labels.
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: Change in z-score
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
Change in z-score | 0.15 (0.77) | 0 (0.73)

5. Secondary Outcome: Facial Affect Recognition (Low Level Social Cognition)
Description: Participants are asked to identify facial expressions of emotion in still photographs from the standardized stimulus set developed by Ekman. The test includes digitized color photos of eight different posers displaying facial expressions of six basic emotions plus neutral expressions. On each trial, a photo and a list of the seven possible expressions are simultaneously presented on the screen. The participant verbally identifies the emotion he/she believes is correct and the experimenter enters the response. The dependent measure is the total number correct.
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: Change in z-score
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
Change in z-score | 0.05 (0.67) | 0.22 (0.45)

6. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) for Schizophrenia Total Score
Description: This is a frequently used instrument, initially developed by Kay, Opler, and Fiszbein, that assesses 30 different symptoms (categorized into positive, negative, and general psychopathology) on a scale from 1 to 7, based on clinical interview. It will be used to compare the psychopathology between the two treatment groups.
  The maximum Total Score on the scale is 210 and the minimum score is 30, with higher values indicating more severe symptoms. The maximum scale of 210 is the sum of the scores from each symptom category (positive symptoms = range 7 to 49; negative symptoms = range 7 to 49; general psychopathology = range to 16 to 112).
  Our outcome measure refers to the change in the PANSS Total Score. A greater decrease on the scale indicates greater improvement in symptoms (e.g., a participant with a change score of -20 improved more on the PANSS than a participant with a change score of -5).
Time Frame: Visit 2 (baseline), Visit 3 (1 week following, post-treatment)
Measure: Mean (Standard Deviation); unit: change in units on scale
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Number analyzed (Participants) | 12 | 11
change in units on scale | -10.83 (5.37) | -8.89 (6.19)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month.
Arm/Group | Inactive Nasal Spray | Intranasal Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 2/12 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inactive Nasal Spray (N=12) | Intranasal Oxytocin (N=11)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Mild rhinorrhea
Mild nasal tingling/irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Mild tingling/irritation after receiving nasal spray
Drowsiness (Nervous system disorders) | 0 | 1 — General drowsiness/sedation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes